CLINICAL TRIAL: NCT01608542
Title: A Phase I, Open-label Study to Assess the Pharmacokinetics of Oral Fostamatinib in Healthy Japanese Subjects After Single and Multiple Doses
Brief Title: A Single and Multiple Dose Study to Assess Blood and Urine Drug Levels of Fostamatinib in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00032
Record Dates: First submitted 2012-05-30; First posted 2012-05-31 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Healthy Japanese Volunteers
Keywords: fostamatinib; FosD; Japanese Healthy volunteers; Phase 1; Single and Multiple Dose Study
MeSH Terms: interventions — fostamatinib

ARMS (2):
- Fostamatinib 100mg (Experimental): Up to two cohorts of Japanese subjects are planned to receive fostamatinib 100mg single and multiple twice daily doses
  Interventions: Drug: Fostamatinib 100mg
- Fostamatinib 200mg (Experimental): Up to two cohorts of Japanese subjects are planned to receive fostamatinib 200mg single and multiple twice daily doses
  Interventions: Drug: Fostamatinib 200mg

INTERVENTIONS:
Drug: Fostamatinib 100mg — oral tablet
  Arms: Fostamatinib 100mg
Drug: Fostamatinib 200mg — oral tablet
  Arms: Fostamatinib 200mg

SUMMARY:
This is a single and multiple dose study in healthy male and female (of non-child bearing potential) Japanese volunteers, to assess the blood and urine drug levels of Fostamatinib. Fostamatinib is being developed for the treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
A Phase I, Open-label Study to Assess the Pharmacokinetics of Oral Fostamatinib in Healthy Japanese Subjects After Single and Multiple Doses

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (of non-childbearing potential) Japanese subjects
* 20 to 45 years of age
* Body mass index (BMI) between 17 and 27 kg/m2 and weigh at least 45 kg and no more than 100 kg

Exclusion Criteria:

* History or presence of respiratory, GI, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders
* Any clinically significant illness, acute infection, known inflammatory process, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product
* Smoking in excess of 5 cigarettes per day or equivalent within 30 days of Day 1
* Use of prescription or over-the-counter drugs within 2 weeks of first administration of investigational product
* Previous participation in a fostamatinib study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of fostamatinib from blood and urine in terms of AUC; tmax; Cmax; t1/2 and Rac. | PK sampling at predose, 0, 0.25, 0.5, 1,1.5, 2, 4, 6, 8,12, 16, 24, 36, 48 and 72 hours post-dose following the single dose (on Day 1) and after repeated twice daily dosing on Days 4 and 10
  AUC - area under the plasma concentration time curve from zero to infinity ; tmax - time to max plasma concentration; t1/2 - terminal elimination half life; Rac - accumulation ratio

SECONDARY OUTCOMES:
Safety and tolerability profile in terms of adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, 12 lead ECG | Up to Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, Study Director — AstraZeneca; David Han, MD, Principal Investigator — PAREXEL Early Phase/California Clinical Trials Medical Group
Locations (2):
- United States (2):
  - Glendale, California
  - Baltimore, Maryland